CLINICAL TRIAL: NCT01061372
Title: Randomized Double-Blind, 12-Week Study Of Pregabalin In Subjects With Restless Legs Syndrome
Brief Title: 12-Week Efficacy And Safety Of Pregabalin In Treating Restless Legs Syndrome (RLS) Subjects
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081184
Record Dates: First submitted 2010-02-01; First posted 2010-02-03 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2010-06

CONDITIONS: Restless Legs Syndrome
Keywords: RLS
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Pregabalin 150 mg/day (Experimental)
  Interventions: Drug: pregabalin
- Pregabalin 300 mg/day (Experimental)
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: Placebo — Placebo, orally administered once a day, 1-3 hours before bedtime for 12 weeks
  Arms: Placebo
Drug: pregabalin — pregabalin 150 mg, orally administered once a day, 1- 3 hours before the bedtime for 12 weeks
  Other Names: Lyrica
  Arms: Pregabalin 150 mg/day
Drug: pregabalin — pregabalin 300 mg, orally administered once a day, 1- 3 hours before the bedtime for 12 weeks
  Other Names: Lyrica
  Arms: Pregabalin 300 mg/day

SUMMARY:
The purpose of this study is to assess efficacy and safety of pregabalin in treating moderate to severe Restless Legs Syndrome in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Restless Legs Syndrome with the presence of all four clinical manifestations of RLS:
* RLS symptoms occur predominantly in the evening
* RLS history at least 6 months
* International Restless Legs Study Group Rating Scale (IRLS) greater than or equal to 15 at the beginning and the end of placebo run-in
* Have greater than or equal to 15 nights with RLS symptoms in the month prior to screening

Exclusion Criteria:

* Any secondary RLS
* Current augmentation due to RLS treatment
* Placebo responders identified during the placebo run-in

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in RLS symptom severity using the International Restless Leg Group Rating Scale (IRLS) total score for efficacy assessment | up to 12 weeks
The proportion of subjects responding to treatment using the Clinical Global Impression - Improvement (CGI-I) scale for efficacy assessment | up to 12 weeks

SECONDARY OUTCOMES:
Subjective Sleep Questionnaire (SSQ - Subjective WASO) | up to 12 weeks
RLS Next Day Impact (RLS-NDI) | up to 12 weeks
Limb pain rating using a numerical rating scale (Limb Pain - NRS) | up to 12 weeks
Clinical Global Impressions - Severity (CGI-S) | up to 12 weeks
Medical Outcomes Study - Sleep Scale (MOS - SS) | up to 12 weeks
Impact on Life (IRLS symptom impact sub-score) | up to 12 weeks
RLS-Quality of Life Scale (RLS-QoL) | up to 12 weeks
Medical Outcomes Study - Short Form 36 (SF-36) | up to 12 weeks
Work Productivity and Activity Impairment - Specific Health Problem (WPAI-SHP) | up to 12 weeks
Profile of Mood States (POMS) | up to 12 weeks
Adverse events from spontaneous reports will be monitored throughout the trial and summarized by treatment group | up to 12 weeks
Sheehan Suicidality Tracking Scale (S-STS) will be utilized to assess the risk of suicide | up to 12 weeks
Changes in RLS symptoms following the discontinuation of study drug at the end of treatment will be evaluated by collection of the IRLS scores at the end of the drug taper period at Week 13 | week 13

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081184&StudyName=12-Week%20Efficacy%20And%20Safety%20Of%20Pregabalin%20In%20Treating%20Restless%20Legs%20Syndrome%20%28RLS%29%20Subjects